CLINICAL TRIAL: NCT00958685
Title: Effect of Enteral Feeding With Ginger Extract in Acute Respiratory Distress Syndrome
Brief Title: Safety Study of Feeding With Ginger Extract in Acute Respiratory Distress Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Zahra Vahdat Shariatpanahi, Faculty of Nutrition Sciences and Food Technology
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INFI-112
Record Dates: First submitted 2009-08-03; First posted 2009-08-13 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2009-08

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ginger extract; ARDS; enteral feeding; mechanical ventilation; ICU
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — ginger extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ginger (Experimental): Study group received 1200 mg of ginger extract and control group 2 gram of coconut oil as placebo
  Interventions: Dietary Supplement: ginger
- placebo (Experimental): Study group received 1200 mg of ginger extract and control group 2 gram of coconut oil as placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: ginger — Study group received 1200 mg of ginger extract and control group 2 gram of coconut oil as placebo
  Other Names: Zingiber officinale
  Arms: ginger
Dietary Supplement: placebo — Study group received 1200 mg of ginger extract and control group 2 gram of coconut oil as placebo
  Other Names: Zingiber officinale
  Arms: placebo

SUMMARY:
An enteral diet supplemented with ginger extract in acute respiratory distress syndrome (ARDS) patients may be beneficial for gas exchange and could decrease duration of mechanical ventilation and length of stay in intensive care unit (ICU).

DETAILED DESCRIPTION:
Rationale: Clinical ARDS occurs primarily as the result of inflammatory injury to the alveoli producing diffuse alveolar damage.

Objective: To evaluate the effects of an enteral diet enriched with ginger extract on inflammatory factors, respiratory profile and outcome of patients with ARDS.

Methods: In this single center, randomized, controlled double blind study, 32 patients with ARDS were randomized to receive a high protein enteral diet enriched with ginger extract or placebo.

Measurements and Main Results: Serum levels of IL-1, IL-6, TNF-α and LTB-4, oxygenation, measured as PaO2/FiO2, static compliance measured on days 0, 5 and 10.

Patients fed enteral diet enriched with ginger extract had significantly lower serum levels of IL-1, IL-6, TNF-α and LTB-4 on days 5 and 10 compared to control group (P<0.05). Significant improvement in oxygenation was observed on day 5 (P=0.02) and 10 (P=0.003) in ginger extract group compared to control group. Static compliance was also increased significantly on day 5 (P=0.01) in ginger extract group compared to control group. A significant difference was found in duration of mechanical ventilation (P0.02) and length of ICU stay (P=0.04) in favor of ginger extract group. We did not find any difference in barotraumas, organ failure and mortality between the study groups.

Conclusions: An enteral diet supplemented with ginger extract in ARDS patients may be beneficial for gas exchange and could decrease duration of mechanical ventilation and length of stay in ICU.

ELIGIBILITY:
Inclusion Criteria:

* Required positive pressure ventilation via endotracheal tube or tracheostomy and were on enteral nutrition support.
* Also they had to have an acute onset of significantly impaired oxygenation with a PaO2 to FiO2 ratio equal or less than 200, bilateral pulmonary infiltrates on frontal chest radiograph and no clinical evidence of left atrial hypertension according to the American-European Consensus Conference on ARDS .
* Patients had to be enrolled within 48 hours of developing these criteria.

Exclusion Criteria:

* Age younger than 18 years
* Participation in other interventional trials in the previous 30 days
* Neurological conditions that could impair weaning from ventilatory support,
* Severe chronic respiratory disease
* Pregnancy
* Lactation
* Active bleeding
* Head trauma
* Intracranial hemorrhage
* Peptic ulcer
* HIV infection
* Food allergy
* Morbid obesity
* Malignancy or other irreversible conditions for which 6 months mortality was estimated to be 50% or more and who were receiving nonsteroidal anti inflammatory drugs or ketoconazole.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
changes in oxygenation, respiratory mechanics and serum inflammatory factors | 21 days
oxygenation | 21 days

SECONDARY OUTCOMES:
the number of organ failure free days, the occurrence of barotraumas, the number of ventilator free days, the number of ICU free days and ICU mortality. | after intervention

CONTACTS AND LOCATIONS:
Overall Officials: zahra vahdat shariatpanahi, MD, Ph.D, Principal Investigator — Faculty of Nutrition Sciences and Food Technology
Locations (1):
- Faculty of Nutrition Sciences and Food Technology, Tehran, Iran